CLINICAL TRIAL: NCT05519072
Title: Use of Prophylactic Antibiotics Prior to OnabotulinumtoxinA Treatment of Overactive Bladder: a Randomized Controlled Trial
Brief Title: Use of Prophylactic Antibiotics Prior to OnabotulinumtoxinA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Atlantic Health System (Other)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Carolyn Botros, Associate Program Director FPMRS Fellowship, Principal Investigator, Atlantic Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1889711-1
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Antibiotic Prophylaxis
Keywords: Antibiotics; Botox; OnabotulinumtoxinA
MeSH Terms: interventions — Nitrofurantoin; Trimethoprim, Sulfamethoxazole Drug Combination; Trimethoprim; Cephalexin; Ciprofloxacin; Amoxicillin-Potassium Clavulanate Combination; Fosfomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antibiotic arm (Experimental): Antibiotics will be administered for 2 days pre-treatment, on the treatment day, and 2 days post-treatment.
  Interventions: Drug: Nitrofurantoin
- No treatment arm (No Intervention): No antibiotics administered.

INTERVENTIONS:
Drug: Nitrofurantoin — For those randomized to the treatment arm, antibiotics will be prescribed at the discretion of the ordering physician. They will be prescribed only in oral form and in accordance with the patient's allergy profile.
  Other Names: Trimethoprim/Sulfamethoxazole; Trimethoprim; Cefalexin; Ciprofloxacin; Augmentin; Fosfomycin
  Arms: Antibiotic arm

SUMMARY:
This study aims to show that lack of antibiotic prophylaxis to those undergoing bladder Botox injections is not significantly inferior to administering prophylaxis. By proving this, the investigators aim to decrease antibiotic use in this setting to combat the growing issue of antibiotic resistance.

Participants will be randomized to antibiotic or no treatment arm. Those randomized to the treatment arm will receive oral antibiotics for 2 days pre-treatment, on the treatment day, and 2 days post-treatment. Participants will return for a follow up appointment approximately 2 weeks after treatment to assess for urinary tract infection (UTI) symptoms. They will be called again at 6 weeks for follow up.

DETAILED DESCRIPTION:
Single-centered, randomized-controlled trial. Participants will be randomized to antibiotic or no treatment arm. All subjects will obtain a urine culture approximately 14 days before the procedure. Those randomized to the treatment arm will receive oral antibiotics at the discretion of physician in accordance to patient's allergies. Antibiotics will be administered for 2 days pre-treatment, on the treatment day, and 2 days post-treatment.

Technique and dose of Botox injection will be at the discretion of the operating physician. Participants will return for a follow up appointment approximately 2 weeks after treatment as is standard, to check a post void residual. They will be called again at 6 weeks for follow up. The investigators will assess for urinary tract infection symptoms, voiding dysfunction, and other adverse events potentially related to the prophylactic antibiotics. Urine cultures will be collected, when possible, to confirm infection for patients developing symptoms.

For the sample size calculation, the investigators assume an alpha (α) value of 0.05 and a power of 80%. The UTI rate after the bladder Botox procedure is 20% (Chapple et al) and the investigators have chosen a δ of 20%. This was chosen because it was the largest amount the investigators found acceptable to presume the no antibiotic group non-inferior. Using these calculations, 64 persons are needed per study arm. With a 10% drop out rate, a total sample size would equal 140 patients total, with 70 per arm.

If participants are found to meet inclusion criteria, they will be contacted by the study team to assess for desired participation in the study. If the patient is agreeable to participate, a phone or in person consent will be obtained and the patient will be randomized. All participants, regardless of study arm, will have a urine culture collected preoperatively, approximately 14 days before procedure. If found to have a UTI, the participants will be treated accordingly. Those in the no antibiotic treatment arm will not receive any antibiotic prophylaxis and will undergo Botox injection. Those in the treatment arm will receive oral antibiotics prescribed at discretion of physician in accordance to participant's allergies.

The primary concern is the development of adverse side effects to antibiotics. Subjects will be monitored throughout the study for these potential adverse events by screening for symptoms. If an event occurs, the PI will be notified immediately. It will also be reported to the Institutional Review Board (IRB) and to all members of the research team.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age ≥ 18
* Patient undergoing bladder Botox treatment

Exclusion Criteria:

* Pregnant and/or breastfeeding
* Contraindication to injection of Botox - hypersensitivity to any botulinum toxin preparation or to any of the components in the formulation, symptomatic urinary retention or post void residual (PVR) > 200 mL, unwillingness or inability to initiate clean intermittent catheterization (CIC) post-treatment if required.
* Contraindication to oral antibiotics - hypersensitivity or allergy
* Inability to take medication by mouth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2024-08-16 (Estimated); Study Completion 2024-08-16 (Estimated)

PRIMARY OUTCOMES:
Urinary tract infections | 2 weeks post-procedure
  Number of participants with urinary tract infections

SECONDARY OUTCOMES:
Urinary tract infections | 6 weeks post-procedure
  Number of participants with urinary tract infections

OTHER OUTCOMES:
Urinary retention and adverse reactions | 6 weeks
  Number of participants with reactions to antibiotics and urinary retention

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Botros, DO, Principal Investigator — Atlantic Health System
Locations (1):
- Atlantic Health, Morristown, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nitti VW, Ginsberg D, Sievert KD, Sussman D, Radomski S, Sand P, De Ridder D, Jenkins B, Magyar A, Chapple C; 191622-096 Investigators. Durable Efficacy and Safety of Long-Term OnabotulinumtoxinA Treatment in Patients with Overactive Bladder Syndrome: Final Results of a 3.5-Year Study. J Urol. 2016 Sep;196(3):791-800. doi: 10.1016/j.juro.2016.03.146. Epub 2016 Mar 30. PMID 27038769
- [Background] Hashim H, Beusterien K, Bridges JF, Amos K, Cardozo L. Patient preferences for treating refractory overactive bladder in the UK. Int Urol Nephrol. 2015 Oct;47(10):1619-27. doi: 10.1007/s11255-015-1100-3. Epub 2015 Sep 7. PMID 26347077
- [Background] Sievert KD, Chapple C, Herschorn S, Joshi M, Zhou J, Nardo C, Nitti VW. OnabotulinumtoxinA 100U provides significant improvements in overactive bladder symptoms in patients with urinary incontinence regardless of the number of anticholinergic therapies used or reason for inadequate management of overactive bladder. Int J Clin Pract. 2014 Oct;68(10):1246-56. doi: 10.1111/ijcp.12443. Epub 2014 Apr 22. PMID 24754838
- [Background] Kuo YC, Kuo HC. Adverse Events of Intravesical OnabotulinumtoxinA Injection between Patients with Overactive Bladder and Interstitial Cystitis--Different Mechanisms of Action of Botox on Bladder Dysfunction? Toxins (Basel). 2016 Mar 16;8(3):75. doi: 10.3390/toxins8030075. PMID 26999201
- [Background] Houman J, Moradzadeh A, Patel DN, Asanad K, Anger JT, Eilber KS. What is the ideal antibiotic prophylaxis for intravesically administered Botox injection? A comparison of two different regimens. Int Urogynecol J. 2019 May;30(5):701-704. doi: 10.1007/s00192-018-3721-4. Epub 2018 Aug 3. PMID 30074062
- [Background] Wencewicz TA. Crossroads of Antibiotic Resistance and Biosynthesis. J Mol Biol. 2019 Aug 23;431(18):3370-3399. doi: 10.1016/j.jmb.2019.06.033. Epub 2019 Jul 6. PMID 31288031
- [Background] Huemer M, Mairpady Shambat S, Brugger SD, Zinkernagel AS. Antibiotic resistance and persistence-Implications for human health and treatment perspectives. EMBO Rep. 2020 Dec 3;21(12):e51034. doi: 10.15252/embr.202051034. Epub 2020 Dec 8. PMID 33400359
- [Background] Eckhardt SE, Takashima Y, Handler SJ, Tenggardjaja C, Yazdany T. Antibiotic regimen and route of administration do not alter rates of urinary tract infection after intravesical botulinum toxin injection for overactive bladder. Int Urogynecol J. 2022 Mar;33(3):703-709. doi: 10.1007/s00192-021-04691-4. Epub 2021 Feb 16. PMID 33594517
- [Background] Lightner DJ, Wymer K, Sanchez J, Kavoussi L. Best Practice Statement on Urologic Procedures and Antimicrobial Prophylaxis. J Urol. 2020 Feb;203(2):351-356. doi: 10.1097/JU.0000000000000509. Epub 2019 Aug 23. PMID 31441676
- [Background] Khan MH, Baldo O, Koenig P, Shaikh N. Use of prophylactic antibiotics for intra-vesicle Botox(R) injection. Neurourol Urodyn. 2017 Mar;36(3):828. doi: 10.1002/nau.23034. Epub 2016 May 13. PMID 27177011
- [Background] Chapple C, Sievert KD, MacDiarmid S, Khullar V, Radziszewski P, Nardo C, Thompson C, Zhou J, Haag-Molkenteller C. OnabotulinumtoxinA 100 U significantly improves all idiopathic overactive bladder symptoms and quality of life in patients with overactive bladder and urinary incontinence: a randomised, double-blind, placebo-controlled trial. Eur Urol. 2013 Aug;64(2):249-56. doi: 10.1016/j.eururo.2013.04.001. Epub 2013 Apr 10. PMID 23608668